CLINICAL TRIAL: NCT04166227
Title: Clinical and Cost-effectiveness of Hip Arthroscopy Versus Definitive Total Hip Arthroplasty in 40-60 Year Olds With Early Hip Osteoarthritis: A Randomized Trial
Brief Title: Hip Arthroscopy Versus Total Hip Arthroplasty RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Ryan Degen, Orthopaedic Surgeon, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114679
Record Dates: First submitted 2019-11-12; First posted 2019-11-18 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Hip Osteoarthritis
Keywords: Hip Scope; Total Hip Replacement
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip Arthroscopy (Active Comparator): Patients in the Hip Arthroscopy group will undergo arthroscopy in the supine position under general anesthesia, with all procedures performed by two subspecialty-trained hip arthroscopists. An algorithmic surgical approach will be utilized to sequentially address pathology in the central and peripheral compartments of the hip based on both preoperative imaging findings and intraoperative findings. Emphasis will be placed on labral preservation and refixation, with osseous decompression under fluoroscopic guidance.
  Interventions: Procedure: Hip Arthroscopy
- Total Hip Arthroplasty (Active Comparator): Patients randomized to the Total Hip Replacement (THR) group will undergo THR via a direct anterior approach. A slightly oblique skin incision measuring approximately 8 cm will be used, starting 3 cm distally and laterally to the anterosuperior iliac spine. The intervals between tensor fascia lata (TFL) and sartorius will be developed superficially, and between rectus femoris and gluteus minimus deeper. Capsulotomy will be performed. A double osteotomy of the femoral neck will be performed to facilitate removal of the head followed by traditional preparation of the acetabulum using an offset reamer and the acetabular component will be inserted. Next, the superior capsule will be released to elevate the femur to allow access to the femoral canal, followed by standard preparation by use of an offset broach and the stem will be implanted
  Interventions: Procedure: Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Hip Arthroscopy — Patients in the Hip Arthroscopy group will undergo arthroscopy in the supine position under general anesthesia, with all procedures performed by two subspecialty-trained hip arthroscopists. An algorithmic surgical approach will be utilized to sequentially address pathology in the central and peripheral compartments of the hip based on both preoperative imaging findings and intraoperative findings. Emphasis will be placed on labral preservation and refixation, with osseous decompression under fluoroscopic guidance.
  Arms: Hip Arthroscopy
Procedure: Total Hip Arthroplasty — Patients randomized to the Total Hip Replacement (THR) group will undergo THR via a direct anterior approach. A slightly oblique skin incision measuring approximately 8 cm will be used, starting 3 cm distally and laterally to the anterosuperior iliac spine. The intervals between tensor fascia lata (TFL) and sartorius will be developed superficially, and between rectus femoris and gluteus minimus deeper. Capsulotomy will be performed. A double osteotomy of the femoral neck will be performed to facilitate removal of the head followed by traditional preparation of the acetabulum using an offset reamer and the acetabular component will be inserted. Next, the superior capsule will be released to elevate the femur to allow access to the femoral canal, followed by standard preparation by use of an offset broach and the stem will be implanted
  Arms: Total Hip Arthroplasty

SUMMARY:
The aim of the proposed study is to perform a comparative pilot, randomized controlled trial of hip arthroscopy versus definitive total hip arthroplasty (THA) for the treatment of early hip osteoarthritis (Tönnis Grade 1-2) in patients between the ages of 40-60 years.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a randomized trial to compare hip arthroscopy to THR and estimate the long-term cost-effectiveness. Specifically, we aim to:

1. Estimate the magnitude of the between-groups difference in the primary outcome (Hip Dysfunction and Osteoarthritis Outcome Score - HOOS);
2. Evaluate the clinical and cost-effectiveness of early definitive THA compared to arthroscopy for early-stage hip OA at 1-year postoperative;
3. Estimate the lifetime cost-effectiveness of arthroscopy vs THA using a Markov model; and
4. Identify imaging and biomechanical predictors of outcomes following hip arthroscopy

ELIGIBILITY:
Inclusion criteria:

1. Between the ages of 40-60 years at the time of surgery.
2. Radiographic evidence of mild to moderate hip OA (Tönnis Gr 0 with MRI chondral wear, Tönnis Gr 1 and 2).
3. Patients must have completed ≥3 months of non-operative management with ongoing symptoms.

Exclusion criteria:

1. Advanced OA, defined as <2 mm joint space (Tönnis Gr 3) or those with acetabular or femoral head cysts.
2. Patients who are pregnant or may become pregnant around the time of surgery.
3. Prior arthroplasty of the contralateral hip.
4. Current or prior hip dysplasia (defined by a lateral centre edge angle of <20 degrees).
5. Acetabular protrusio or coxa profunda, making arthroscopic access unsafe/unfeasible.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hip Dysfunction and Osteoarthritis Outcome Score (HOOS) | 6 weeks, 3, 6 and 12 months
  Subscales measuring Pain, Symptoms, Activity limitations daily living and Function in sport and recreation The outcome measure is transformed in a worst to best scale from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms.

SECONDARY OUTCOMES:
Change in International Hip Outcome Tool [iHOT] | 6 weeks, 3, 6 and 12 months
  The iHOT-33 is a validated, self-administered quality of life assessment tool for young, active patients with hip symptoms. Each question is scored from 0-100 and the average for all questions is calculated, where 100 represents the best possible outcome or highest level of function.
Change in Hip Outcome Score | 6 weeks, 3, 6 and 12 months
  Validated measure of hip function, includes subscale of ADL (activities of daily living) and Sport will be utilized. Each HOS subscale is calculated from 0 to 100, with 100 being the best score
Change in Modified Harris Hip Score | 6 weeks, 3, 6 and 12 months
  Min: 0 Max: 100
  Scoring of mHHS:
  Excellent: 90--100 Good: 80--89 Fair: 70--79 Poor: <70
  Higher score indicates better hip functionally.
EQ-5D | 6 weeks, 3, 6 and 12 months
  Health-related quality of life tool to estimate utility scores for the economic analyses (mixed quantitative and qualitative tool with VAS score from 0-100, where 100 represents the 'best imaginable health state')
Cost Utilization | 6 weeks, 3, 6 and 12 months
  Record all procedural related costs for each intervention and any additional direct and indirect resource use over the study period
Magnetic Resonance Imaging (MRI) | Baseline and 12 months
  To enable quantification of morphological features of the hip joint (alpha angle - measured on the axial images; lateral center edge angle measured on the coronal images) and chondral degeneration (Outerbridge classification 0-5)
Change in performance on 40 meter fast-paced walk test | 6 weeks, 3, 6 and 12 months
  Walk as quickly but as safely as possible, without running, along a 10 m (33 ft) walkway and then turn around a cone, return then repeat again for a total distance of 40 m (132 ft) (3 turns). Time is recorded to the nearest 100th second, and speed is then calculated as a value of meters/second.
Change in 6-minute Walk Test | 6 weeks, 3, 6 and 12 months
  Walking from end to end over a premeasured distance, covering as much ground as possible at a comfortable, safe pace. Distance covered in 6 minutes is recorded to the nearest 10th of a meter.
Change in Timed Up and Go Test | 6 weeks, 3, 6 and 12 months
  Starting in a seated position in a standard arm chair (height of 44 cm), the time it takes to stand up, walk 3 meters and return to a seated position. Time is recorded to the nearest 100th of a second.
Change in performance on 30-second Chair Stand Test | 6 weeks, 3, 6 and 12 months
  From the sitting position, stand up completely so hips and knees are fully extended, then completely back down, so that the bottom fully touches the seat. This is repeated as many times as possible in 30 seconds. Score is the total number of completed repetitions.
3-dimensional gait analysis to provide walking characteristics (gait velocity, step length, stride length), kinematics (hip joint angles, pelvic tilt, lateral trunk lean) and kinetics (hip joint moments) | 6 weeks, 3, 6 and 12 months
  12-camera, motion capture system, and a synchronized floor-mounted force platform will be used. Passive-reflective markers are placed on patients using a 22-marker, modified Helen Hayes marker set. Patients will be instructed to walk barefoot across an 8-m walkway at their typical self-selected walking speed, until at least five successful force plates strikes are collected for each limb. Three-dimensional joint angles and moments are calculated from the kinematic and kinetic data using commercial software (Orthotrak 6.6; Motion Analysis Corporation, Santa Rosa, CA) and custom post processing and data reduction techniques

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Degen, MD, FRCSC, Principal Investigator — Fowler Kennedy Sport Medicine Clinic
Locations (2):
- Canada (2):
  - Fraser Health, New Westminster, British Columbia
  - Fowler Kennedy Sport Medicine Clinic and University Hospital, London, Ontario